CLINICAL TRIAL: NCT01154842
Title: Serum Fibroblast Growth Factor-23 (FGF-23) Levels Are Independently Associated With Left Ventricular Mass and Myocardial Performance Index in Maintenance Haemodialysis Patients
Brief Title: Fibroblast Growth Factor-23 (FGF-23) is Independently Associated With Left Ventricular Mass Index (LVMI) and Myocardial Performance Index (MPI) in Haemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Diskapi Training and Research Hospital, Diskapi Training and Research Hospital
Other Study IDs: 1-perk
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-01

CONDITIONS: Fibroblast
Keywords: FGF-23; Dialysis; plasma FGF-23 levels; echocardiography

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human plasma to measure FGF-23 levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis: Adult hemodialysis patients (age>18 years)

SUMMARY:
Serum FGF-23 levels will be measured in patients with a history of coronary artery disease and aortic valve calcifications.It will be searched whether patients with MPI>0.47 had higher or lower serum FGF-23 levels than those with MPI<0.47. Correlations will be examined between log FGF-23 levels and LVMI and MPI. Uni and Multivariable-adjusted regression analyses regarding whether increased log FGF-23 concentrations are independently associated with increased left ventricular mass index and increased MPI, will be performed.

DETAILED DESCRIPTION:
Fibroblast growth factor 23 (FGF-23) is a phosphorus-regulating substance. Circulating FGF-23 levels increase markedly in dialysis patients and are independently associated with increased risk of mortality. Given the fact that cardiovascular disease is the leading cause of death in dialysis patients, the aim of this study was to test if elevated FGF-23 levels might be associated with left ventricular mass index (LVMI) and left ventricular index of myocardial performance (MPI) in maintenance haemodialysis patients.

Methods: In this cross-sectional study, plasma FGF-23 concentrations are measured using a C-terminal human enzyme-linked immunosorbent assay kit and echocardiography is performed in maintenance haemodialysis patients.

Serum FGF-23 levels will be measured in patients with a history of coronary artery disease and aortic valve calcifications.It will be searched whether patients with MPI>0.47 had higher or lower serum FGF-23 levels than those with MPI<0.47. Correlations will be examined between log FGF-23 levels and LVMI and MPI. Uni and Multivariable-adjusted regression analyses regarding whether increased log FGF-23 concentrations are independently associated with increased left ventricular mass index and increased MPI, will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients (age>18 years old)

Exclusion Criteria:

* Malignancy, active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hemodialysis patients (age>18 years old)
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To test if elevated FGF-23 levels might be associated with left ventricular mass index (LVMI) and left ventricular index of myocardial performance (MPI) in maintenance haemodialysis patients. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: ALPER KIRKPANTUR, Assoc Prof, Study Chair — Diskapi Training and Research Hospital; MUSTAFA BALCI, Dr, Study Chair — Diskapi Training and Research Hospital; OGUZ GURBUZ, Dr, Study Chair — Diskapi Training and Research Hospital; BARIS AFSAR, Dr, Study Chair — Zonguldak Training and Research Hospital; BASOL CANBAKAN, Assoc Prof, Study Chair — Diskapi Training and Research Hospital; RAMAZAN AKDEMIR, Assoc Prof, Study Chair — Diskapi Training and Research Hospital; DENIZ AYLI, Assoc Prof, Study Director — Diskapi Training and Research Hospital
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)